CLINICAL TRIAL: NCT07326930
Title: Tracjectories and Predictors of Chemotherapy Induced Peripheral Neuropathy in Children With Acute Lymphoblastic Leukemia: A Perspective Longitudinal Study
Brief Title: Tracjectories and Predictors of Chemotherapy Induced Peripheral Neuropathy in Children With Acute Lymphoblastic Leukemia
Status: Recruiting | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Eva Ho, Associate professor, The Hong Kong Polytechnic University
Other Study IDs: CIPN trajectories
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphoblastic Leukemia ALL
Keywords: Chemotherapy induced peripheral neuropathy; tracjectory; predictor; children; acute lymphoblastic leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire: Participants will complete chemotherapy induced peripheral neuropathy, physical symptoms, nutrition status, psychological distress, sleep quality, physical activity, perceived social support and coping strategy scales.

SUMMARY:
The goal of this study is to explore the trajectory patterns of chemotherapy induced peripheral neuropathy over the course of chemotherapy and identify predictors of distinct trajectories in children with acute lymphoblastic leukemia. A perspective longitudinal study design is utilized. Chemotherapy induced peripheral neuropathy was assessed at one week after the first use of Vincristine (VCR) (T1), one week after the second use of VCR (T2), one week after the third use of VCR (T3), one week after the fourth use of VCR (T4), two weeks after T4 (T5), two weeks after T5 (T6), two weeks after T5 (T7). Patients' demographic and clinical characteristics, physical symptoms, nutrition status, psychological distress, sleep quality, physical activity, perceived social support and coping strategy are obtained at baseline.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with acute lymphoblastic leukemia
* aged from 8 to 17 years
* will receive vincristine according the Chinese Children's Cancer Group Acute Lymphoblastic Leukemia-2020 Project (CCCG-ALL-2020)
* conscious with sufficient cognitive abilities to understand and express their physical state and psychological feelings accurately
* written informed assent is obtained from the children and their parents for their participation in the study

Exclusion Criteria:

* participating other experimental trials, such as electrical stimulation, exercise therapy may improve CIPN symptoms.
* with severe complications, including but not limited to significant heart, brain, or lung function failure.
* had peripheral neuropathy symptoms caused by other diseases like genetic diseases, spinal cord injury.
* had neuromuscular diseases (e.g., traumatic brain injury and cerebral palsy).
* had central nervous system cancer or secondary cancer.
* had multiple treatment like radiotherapy.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with acute lymphoblastic leukemia are recruited from inpatient wards in Shenzhen Children's Hospital, Henan Cancer Hospital and Shanghai Children's Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-01-07 (Estimated); Study Completion 2026-01-07 (Estimated)

PRIMARY OUTCOMES:
Pediatric chemotherapy-induced peripheral neuropathy (P-CIN) scale | One week after the first use of Vincristine (VCR) (T1), one week after the second use of VCR (T2), one week after the third use of VCR (T3), one week after the fourth use of VCR (T4), two weeks after T4(T5), two weeks after T5(T6), two weeks after T6(T7)
  For measuring participants' peripheral neuropathy induced by chemotherapy. The total score ranges from 0 to 65 with higher scores indicating more severe chemotherpay induced peripheral neuropathy.

OTHER OUTCOMES:
The therapy-related symptom checklist for children (TRSC-C) | Baseline
  TRSC-C is used to assess the participants' physcial symptoms. This checklist contains 30 items divided into 7 factors (1) nutrition-related, (2) psychosocial/ central nervous system (CNS), (3) oropharyngeal, (4) bone marrow toxicity/neuropathy, (5) skin/other toxicities, (6) neurotoxicities, and (7) respiratory/other symptoms. The total TRSC-C score is computed as the average of the symptom scores for all 30 symptoms. Higher scores indicating greater severity of symptoms
Screening tool for the assessment of malnutrition in pediatrics, STAMP | Baseline
  The STAMP is used to assess the nutritional status of participants. The nutritional risk is divided into low risk (0-1 points), moderate risk (2-3 points), and high risk (≥4 points) based on the total score (0-9 points).
National Comprehensive Cancer Network (NCCN) distress thermometer (DT) | Baseline
  The NCCN-DT was used to assess psychological distress among participants. A cut off value ≥4 for single-item DT screening tool is recommended to indicate a distressed patient.
A specific item - 'subjective sleep quality' from the Pittsburgh Sleep Quality Index scale, PSQI | Baseline
  A specific item - 'subjective sleep quality' from PSQI is used to assess the participants' sleep quality. Answer is coded into a 0-3 score for this item, with higher score reflect poor sleep quality.
Leisure Score Index (LSI) of the Godin-Leisure-Time Exercise Questionnaire (GLTEQ) | Baseline
  Leisure Score Index is used to assess the participants' physical activity level. A score of 24 or over indicate active physical activity and higher scores indicating higher levels of physical activity.
Multidimensional Scale of Perceived Social Support, MSPSS | Baseline
  MSPSS is used to assess the participants' perceived social support. The total score ranges from 12 to 84, with higher mean score indicate greater level of Perceived Social Support.
Paediatric Cancer Coping Scale, PCCS | Baseline
  PCCS is used to assess the participants' coping strategies. This scale is divided into three domains: cognitive coping (14 items), problem-oriented coping (9 items) and defensive coping (10 items) with total 33 items. Each item is performed on a 4-point Likert scale from 0 (never) to 3 (always), with higher scores indicating the most frequently used coping strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Ka Yan Ho, Principal Investigator — The Hong Kong Polytechnic University
Locations (3):
- China (3):
  - The Affiliated Cancer Hospital of Zhengzhou University, Henan Cancer Hospital,, Zhengzhou, Henan
  - Shanghai Children's Medical Center, Shanghai
  - Shenzhen Children's Hospital, Shenzhen

IPD SHARING:
Plan to Share IPD: No